CLINICAL TRIAL: NCT06047392
Title: A Pilot Clinical Trial of CT Coronary Angiography for Patients With Suspected Type 2 Myocardial Infarction
Brief Title: CT Coronary Angiography for Type 2 Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GN22CA430
Record Dates: First submitted 2023-08-02; First posted 2023-09-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: Computed Tomography; Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention)
- CT coronary angiography + usual care (Active Comparator)
  Interventions: Diagnostic Test: CT coronary angiography

INTERVENTIONS:
Diagnostic Test: CT coronary angiography — Patients will undergo a CTCA according to local, standard protocol.
  Arms: CT coronary angiography + usual care

SUMMARY:
This study is to explore whether a computed tomography (CT) scan of the heart arteries might improve the care of patients that have presented with a suspected Type 2 myocardial infarction (MI). The Investigators hope to demonstrate that these patients may be the ideal group of patients to benefit from cardiac CT scan imaging by; 1. confirming whether they have any disease in their heart arteries 2. demonstrating the severity of the heart artery disease 3. revealing an alternative cause for their presentation 4. avoiding the need for an invasive heart artery angiogram.

DETAILED DESCRIPTION:
An increasing number of patients present to hospital with a heart attack (myocardial infarction, MI). Heart attacks can be caused by instability and narrowing in heart arteries (Type 1 MI) or strain on the heart (Type 2 MI). Type 2 MIs can be the result of other problems with the heart including inflammation and rhythm problems or other conditions such as infection or low blood count. Both Type 1 and Type 2 MI patients have increased risk of further problems following this presentation. Deciding whether a patient has suffered a Type 1 MI or a Type 2 MI can be very difficult leaving uncertainty for patients and health care staff. Often patients with Type 2 myocardial infarction are either referred for an invasive coronary angiogram (a procedure where dye is injected into the heart arteries directly) or have no further investigations. Invasive angiograms carry a small risk of complications including heart attack, stroke and, rarely, death.

Cardiac CT scanning has emerged in the last 20 years as the first test usually performed to investigate patients that present with stable chest pain symptoms to the outpatient department. The role of cardiac CT in patients that present as an emergency with a suspected heart attack is not yet established.

To date, there are no substantive data on the role of computed tomography coronary angiography (CTCA) in patients with known or suspected Type 2 MI. A pilot study is proposed to address the information gaps. The specific areas of uncertainty include feasibility of enrolling into an imaging trial during acute medical care, feasibility of randomisation (including compliance and cross-overs), incremental diagnostic value, safety (procedure and post-procedure) and healthcare resource utilisation. The study aims to address the gap in evidence highlighted by the recent European Society of Cardiology Guidelines for the management of acute coronary syndromes, 'evaluating diagnostic strategies to better classify patients according to their type of MI (Type 1 vs Type 2)'.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected Type 2 MI

Exclusion Criteria:

1. Unable to provide written informed consent
2. Known severe coronary artery disease
3. Previous PCI
4. Previous CABG
5. Severe renal dysfunction, defined as an eGFR <30 mL/min/1.73 m2
6. Tachycardia (>75bpm) refractory to heart rate control
7. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in primary diagnosis | At discharge from recruiting hospital (assessed up to day 30)
  The primary outcome is a change in the primary diagnosis defined as a difference in the final diagnosis at discharge compared to the initial diagnosis prior to study recruitment. The primary outcome will therefore take account of the diagnostic effect of CTCA and any changes that might normally occur during standard care.

SECONDARY OUTCOMES:
Rate of invasive coronary angiography | 3 months
  Patients undergoing invasive coronary angiography following presentation
Major adverse cardiovascular events | 12 months
  Myocardial infarction, stroke or death
Rate of coronary revascularisation | 12 months
  Either percutaneous coronary intervention or coronary artery bypass grafting
Rate of hospital readmission | 12 months
  Readmission to hospital for any reason
Rate of additional cardiovascular investigations | 12 months
  Referral to outpatient clinic or for additional cardiovascular test (including exercise tolerance testing, echocardiography, myocardial perfusion imaging, cardiac MRI)
Health related quality of life assessment | 6 months
  EQ-5D-5L questionnaire. Reported as 5 digit code (Range 11111 - 55555) with higher numbers indicating worse quality of life and EQ visual analogue scale (Range 0-100) with higher numbers indicating better quality of life.
Functional assessment | 6 months
  Duke Activity Status Index (DASI). Range 0 - 58.2. Higher score indicates better functional status.
Estimated cost of health care | 12 months
  Health care resource utilisation including length of hospital stay, investigations and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Good, MD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J Acute Cardiovasc Care. 2024 Feb 9;13(1):55-161. doi: 10.1093/ehjacc/zuad107. No abstract available. PMID 37740496